CLINICAL TRIAL: NCT04682652
Title: GRAVITY: Genicular Artery Embolization Versus Observation for the Treatment of Symptomatic Knee Osteoarthritis: a Randomized Controlled Trial
Brief Title: Genicular Artery Embolization Vs Observation for Symptomatic Knee Osteoarthritis
Acronym: GRAVITY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Siddharth Padia, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22-001004
Record Dates: First submitted 2020-12-14; First posted 2020-12-24 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis; Degenerative Joint Disease of Knee
Keywords: Microspheres; Artery Embolization; Knee Osteoarthritis; Chronic Pain; Embozene
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain | interventions — Microspheres; Embolization, Therapeutic

STUDY DESIGN:
Intervention Model Description: A total of 100 subjects will be enrolled in the double-arm study, subjects will be randomized to GAE or observation in a 2:1 ratio (67 assigned to GAE, 33 assigned to observational). Subjects in the observation group will have the option to crossover to the GAE treatment arm after they've completed their 6-month follow-up time point. Subjects who crossover to treatment arm will undergo the GAE procedure and undergo all subsequent follow-up visits (1 month, 3 month, 6 month, 12 month, 24 month).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- GAE Treatment (Experimental): Subjects will be treated with a genicular artery embolization (GAE) procedure performed with Embozene Microspheres. The microspheres will be delivered in a saline-contrast medium solution and will be delivered to the arteries supplying the areas of the subject's pain.
  Interventions: Device: Embozene MicroSpheres
- Observational (No Intervention): Subjects randomized to the observational group will not undergo the experimental GAE Treatment.
  PI will offer subjects enrolled into the observational group to crossover to the experimental GAE Treatment group after they have completed their 6-month follow-up assessments.

INTERVENTIONS:
Device: Embozene MicroSpheres — Embozene is a medical device made by Boston Scientific approved in the United States for the treatment of hypervascular tumors and arteriovenous malformations. It consists of thousands of microscopic spheres that are injected into the artery in the knee going to the region of pain. One of the causes of pain in the setting of knee arthritis is increased blood flow going to the specific area of pain. The goal of this procedure is to decrease the blood flow (embolize) to the specific region of the knee that is causing your pain. This is done by infusing Embozene particles into the specific blood vessel (genicular artery) supplying the area of pain in the knee.
  Other Names: Color-Advanced Microspheres; Microspheres for Embolization
  Arms: GAE Treatment

SUMMARY:
The purpose of this clinical trial is to determine whether genicular artery embolization (GAE) is an effective way to treat knee pain from osteoarthritis. Pain from arthritis is often due to underlying inflammation in the joint. The inflammation is associated with increased abnormal blood flow going to the specific area of pain. If the investigator can reduce the blood flow, the inflammation can be reduced and the pain can be controlled.

The GAE procedure is an experimental procedure to decrease the blood flow (embolize) to the specific region of the knee that is causing the pain. This will be done by infusing microscopic spheres into the specific blood vessel (genicular artery) supplying the area of pain in the knee. This is done through a procedure which is called an angiogram, which is done entirely through a pinhole at the creased of the thigh, using twilight (conscious) sedation.

The investigators have already completed an initial trial at UCLA, and shown that this procedure is safe and effective. The purpose of this new trial is to compare outcomes of people undergoing the GAE procedure to those who do not undergo the procedure. A total of 100 patients will be enrolled, and 2/3 of the patients will be randomly selected to undergo the GAE procedure. 1/3 will not undergo the procedure. This is known as a randomized trial. During the trial, all subjects will also get MRIs and fluid withdrawn from their knee joints at various timepoints in order to precisely figure out how the procedure works on a closer (microscopic) level.

DETAILED DESCRIPTION:
This is a single-center, prospective, open-label randomized trial to compare outcomes of GAE versus observation, and to identify biomarkers and imaging endpoints that change in response to GAE.

Subjects will be considered enrolled in the study once they have provided informed consent and have been determined to meet all eligibility criteria. A total of 100 subjects will be enrolled in the double-arm study and will be followed for 24 months.

The study will involve a screening period in which patient eligibility is determined. Once eligibility is confirmed, subjects will then be randomized to GAE or observation in a 2:1 ratio. Group sample sizes of 67 and 33 achieve approximately 85% power to reject the null hypothesis of no difference in the clinical response defined by 50% or greater reduction in WOMAC between the treatment and observation arms with a significance level (alpha) of 0.050 using a two-sided two-proportions using Fisher's exact test. With 100 symptomatic knee osteoarthritis subjects, the power of study is approximately 85% where we assume a target response rate of 67.5% for the experimental arm and 31% for the observational arm with up to 20% drop-out rate prior to 6 months. All study subjects will undergo the initial procedures, consisting of a history and physical exam, dynamic contrast-enhanced knee MRI, blood serum and joint aspiration with biochemical analysis.

For the treatment arm, subjects will undergo GAE with Embozene microspheres (100 micron) (Varian Medical Systems). Observation group will not receive the GAE procedure at baseline, and will be counseled on conservative management with a referral or prescription for physical therapy. Follow-up visits will be at 1 month (± 2 weeks), 3 months (± 2 weeks), 6 months (± 2 weeks), 12 months (± 2 weeks), and 24 months (± 2 weeks) post-procedure. At these visits, subjects will complete the WOMAC, KOOS5, visual analog scale (VAS) pain score, undergo a directed physical examination, and report any new adverse events (AEs). At 6 and 24 months of follow-up, all subjects will also undergo dynamic contrast-enhanced knee MRI, and serum and joint aspiration with biochemical analysis.

At 6 months, subjects in the observation group will have the option to crossover to the GAE treatment arm. Subjects in the crossover group will then undergo GAE, with follow up at 1 month (± 2 weeks), 3 months (± 2 weeks), 6 months (± 2 weeks), 12 months (± 2 weeks), and 24 months (± 2 weeks) post-GAE. For the purposes of data analyses, the follow-up evaluations for crossover subjects will match those of the initial GAE subjects. For example, if a subject in the observation arm undergoes GAE crossover at 6 months, that will be considered the treatment visit, and then subject will undergo evaluation at 1, 3, 6, 12, and 24 months after GAE.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following inclusion criteria in order to be eligible for this study:

* Provided informed consent
* Age ≥ 40 years and less than 80 years
* Ineligibility for or refusal of surgical management
* Moderate-severe knee pain as determined by visual analog scale > 5 out of 10
* Osteoarthritis based on X-ray. Kellgren-Lawrence score > 2 based on radiograph completed within 3 months of procedure date.
* Resistant/failed conservative treatment (e.g. NSAIDS/physical therapy/steroid joint injection/ hyaluronic acid joint injection) for at least 3 months
* Able to comply with all treatments and protocol follow-up visits

Exclusion Criteria

Subjects that meet any of the following exclusion criteria will not be eligible for this study:

* Mild knee pain as determined by visual analog scale < 5 out of 10
* OA on knee radiograph resulting in greater than 20 degree varus or valgus angulation
* Moderate loss of kidney function, define as estimated glomerular filtration rate of less than 45 mL/min.
* Significant arterial atherosclerosis that would limit selective angiography
* History of fibromyalgia, autoimmune, or inflammatory disorder
* History of any lumbar spine surgery, spine injections, or radicular pain in the extremity believed to originate from the spine
* Allergy to iodinated contrast agents
* Active Infection or malignancy
* Recent (within 12 months) or active cigarette use
* Prior total or partial knee replacement in the subject knee
* Active pregnancy
* Uncorrectable bleeding diasthesis

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes in clinical response | 6 months
  The primary evaluation is the change in clinical response, measured by The Western Ontario and McMaster Universities Arthritis Index (WOMAC). The primary endpoint is percentage of subjects achieving at least a 50% reduction in WOMAC at 6 months with an intent-to-treat analysis.

SECONDARY OUTCOMES:
Short term clinical outcomes | 1 and 3 months
  • Compare clinical success rates (defined as at least 50% reduction in WOMAC) between GAE and observation at 1 and 3 months. This will be a intent-to-treat analysis.
Clinic outcomes at multiple timepoints | 1-24 months
  • Compare clinical success rates (defined as at least 50% reduction in WOMAC) between GAE and observation at various timepoints: 1 months, 3 months, 6 months, 12 months, 24 months. This will be a per-protocol analysis.
Degree of change in clinical outcomes via WOMAC | 1-24 months
  • Compare median decrease in WOMAC (measured by percentage) between GAE and observation at various timepoints: 1 month, 3 months, 6 months, 12 months, 24 months. This will be a per-protocol analysis.
Decrease in pain | 1-24 months
  • Compare median decrease in pain (measured by VAS: visual analog scale) between GAE and observation at various timepoints: 1 month, 3 months, 6 months, 12 months, 24 months. This will be a per-protocol analysis.
Change in quality of life | 1-24 months
  • Compare median improvement in health-related quality of life (measured by KOOS5) between GAE and observation at various timepoints: 1 month, 3 months, 6 months, 12 months, 24 months. This will be a per-protocol analysis.
Change in MRI | 6-24 months
  • To assess changes in imaging (MRI) in patients undergoing GAE versus observation, at 0, 6, and 24 months. This will be a per-protocol exploratory analysis.
Change in inflammatory biomarkers | 6-24 months
  • To assess changes in inflammatory markers in patients undergoing GAE versus observation at 0, 6 and 24 months. This will be a per-protocol exploratory analysis.
Correlation of baseline characteristics with clinical response | 1-24 months
  • To assess how differences in baseline clinical, imaging, and biochemical characteristics correlate with clinical response. This will be a per-protocol exploratory analysis.
Degree of progression of osteoarthritis | 24 months
  • To assess the degree of progression of osteoarthritis via changes in knee radiograph at 0 and 24 months in patients undergoing GAE versus observation. This will be a per-protocol exploratory analysis.
Safety assessment | 24 months
  Assess safety via tabulation of adverse events
Pain medication use | 24 months
  To assess change in pain medication use after GAE versus observation.

CONTACTS AND LOCATIONS:
Overall Officials: Siddharth A Padia, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Santa Monica Hospital, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Padia SA, Genshaft S, Blumstein G, Plotnik A, Kim GHJ, Gilbert SJ, Lauko K, Stavrakis AI. Genicular Artery Embolization for the Treatment of Symptomatic Knee Osteoarthritis. JB JS Open Access. 2021 Oct 21;6(4):e21.00085. doi: 10.2106/JBJS.OA.21.00085. eCollection 2021 Oct-Dec. PMID 34703964